CLINICAL TRIAL: NCT04034524
Title: An Observational Study of Glycemic Control and Cardiovascular Outcomes Among Patients With Type 2 Diabetes Newly Initiating Glucagon-like Peptide-1 Receptor Agonists (GLP1) Versus Basal Insulin in Routine Care Settings
Brief Title: Cardiovascular Outcomes and HbA1c Among Patients With Type 2 Diabetes Newly Initiating GLP1RAs vs Basal Insulin
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Jing Luo, Instructor of Medicine, Brigham and Women's Hospital
Other Study IDs: 2011P002580-118
Record Dates: First submitted 2019-07-24; First posted 2019-07-26 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- New users of GLP1 receptor agonists (exposure)
  Interventions: Drug: GLP-1 receptor agonist
- New users of basal insulin (reference)
  Interventions: Drug: Insulin

INTERVENTIONS:
Drug: GLP-1 receptor agonist — any GLP-1 receptor agonist (other than Saxenda or liraglutide 3.0mg)
  Groups: New users of GLP1 receptor agonists (exposure)
Drug: Insulin — glargine, detemir, neutral protamine Hagedorn (NPH), degludec
  Other Names: Basal Insulin
  Groups: New users of basal insulin (reference)

SUMMARY:
This study will compare hemoglobin a1c (HbA1c) and cardiovascular (CV) outcomes among patients with type 2 diabetes newly initiating a GLP1-receptor agonist or basal insulin.

DETAILED DESCRIPTION:
The 2019 ADA-EASD clinical treatment guidelines recommend a GLP-1RA over basal insulin for patients with type 2 diabetes with suboptimal glycemic control despite metformin and a second-line glucose lowering agent. The basis of this recommendation is due to the side effect profiles of these two medications (i.e. reduced risk of hypoglycemia, some weight loss with GLP-1RA), convenience (once weekly injection) and the fact that the price of insulin has skyrocketed in recent years. Prior head-to-head randomized trials (EAGLE, LEAD 5) comparing select GLP-1RA and basal insulin have found mixed results. In EAGLE, adding either insulin glargine or liraglutide to patients with poorly controlled type 2 diabetes found no differences in the primary outcome (percentage of people reaching HbA1c < 7%). In LEAD 5, liraglutide was associated with a slightly greater HbA1c reduction than glargine, however the dose of insulin was approximately 50% less than the dose used in EAGLE. The objective of this observational study is to describe the comparative effectiveness and safety of newly initiating a GLP1RA versus basal insulin in patients with type 2 diabetes using metformin and another oral glucose lowering medicine.

ELIGIBILITY:
Inclusion Criteria:

* Age>=18 years
* at least 180 days of continuous enrollment prior to index date
* at least 1 Type 2 diabetes diagnosis code prior to index date
* (for cohort #1) at least 2 metformin dispensings prior to index date AND days supply overlap on cohort entry date (with 14 days of grace period before)

Exclusion Criteria:

* any type 1 diabetes diagnosis code prior to index date
* medullary thyroid carcinoma, multiple endocrine neoplasia type 2 (both black box warnings) prior to index date
* h/o pancreatitis
* h/o recurrent hypoglycemia (i.e. more than 1 hospitalization / emergency department encounter in primary diagnosis position for hypoglycemia)
* index injectable is a combination of GLP1-RA plus insulin
* index GLP1-RA is Saxenda (indicated for weight loss) or liraglutide at 3.0mg dose
* index insulin regimen includes both basal and prandial insulin, or premixed insulin
* Any prior GLP1-RA use (Applied washout for 180 days)
* Any prior insulin use; Sometimes insulin is transiently used at diagnosis (Applied washout for 180 days)
* Secondary diabetes
* Gestational diabetes
* Nursing home admission (because we don't have pharmacy claims)
* Age <18 years
* Chronic kidney disease stage 4-6
* Advanced cancer
* End stage renal disease

For A1c cohort only:

-HbA1c >12%

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with type 2 diabetes with prior and concomitant use of metformin and other oral anti diabetic agents
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Time until first composite CV event (myocardial infarction, stroke) | Through Study Completion, an estimated average of 1 year

SECONDARY OUTCOMES:
Time until first myocardial infarction | Through Study Completion, an estimated average of 1 year
Time until first stroke | Through Study Completion, an estimated average of 1 year
Time until first serious hypoglycemic event | Through Study Completion, an estimated average of 1 year
Time until first episode of acute pancreatitis | Through Study Completion, an estimated average of 1 year
Time until first episode of acute cholecystitis | Through Study Completion, an estimated average of 1 year

OTHER OUTCOMES:
Proportion of patients with HbA1c post-index < 7% (EAGLE) | 24 weeks
Proportion of patients with HbA1c post-index < 8% (EAGLE) | 24 weeks
Change from baseline HbA1c | 24 weeks
  Weighted mean

CONTACTS AND LOCATIONS:
Overall Officials: Jessica M Franklin, PHD, Study Chair — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States